CLINICAL TRIAL: NCT07303777
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy, Safety, and Population Pharmacokinetics (PopPK) Profile of ABP-745 in Patients With Atherosclerosis
Brief Title: Efficacy, Safety, and PopPK Profile of ABP-745 in Patients With Atherosclerosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABP-745-202
Record Dates: First submitted 2025-12-23; First posted 2025-12-26 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Atherosclerosis Cardiovascular Disease; ASCVD; ASCVD Management
Keywords: ASCVD; ABP-745

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo group (Placebo Comparator): Existing lipid-lowering maintenance medications unchanged.
  Interventions: Drug: Placebo
- ABP-745 Dose A (Experimental): Existing lipid-lowering maintenance medications unchanged.
  Interventions: Drug: ABP-745 Dose A
- ABP-745 Dose B (Experimental): Existing lipid-lowering maintenance medications unchanged.
  Interventions: Drug: ABP-745 Dose B
- ABP-745 Dose C (Experimental): Existing lipid-lowering maintenance medications unchanged.
  Interventions: Drug: ABP-745 Dose C

INTERVENTIONS:
Drug: ABP-745 Dose A — ABP-745 Dose A - tablets (PO), low dose , QD
  Arms: ABP-745 Dose A
Drug: Placebo — ABP-745 placebo - tablets (PO), non-active,QD
  Arms: Placebo group
Drug: ABP-745 Dose B — ABP-745 Dose B - tablets (PO), Midum dose, QD
  Arms: ABP-745 Dose B
Drug: ABP-745 Dose C — ABP-745 Dose C - tablets (PO), High dose, QD
  Arms: ABP-745 Dose C

SUMMARY:
This is a multicenter, randomized, double-blind, placebo parallel controlled study to evaluate the preliminary efficacy, safety, and PopPK profile of ABP-745 in patients with ASCVD. Efficacy of ABP-745 in reducing atherosclerotic plaque compared with placebo will be evaluated in participants with ASCVD. The primary efficacy measurement will be assessed at 52W of treatment.

ELIGIBILITY:
Inclusion Criteria:

Unless otherwise specified, subjects must meet all of the following criteria at screening:

* Diagnosed with coronary at herosclerosis, and coronary angiography.
* Male or female at 18-75 years of age (inclusive).
* Weight ≥40 kg.
* Currently using any oral lipid-lowering therapy.
* Able to understand and willing to sign an ICF and comply with study requirements.
* A woman or man of childbearing potential agreeing to use medically approved contraceptive methods from the screening until 3 months after the last study dose.

Exclusion Criteria:

Unless otherwise specified, subjects are excluded from the study if any of the following criteria is met:

* History of stroke within the past 6 months.
* Uncontrolled arrhythmia within 3 months prior to screening.
* Evidence of any active or suspected cancer within 3 years prior to the screening.
* Having undergone any major surgery within 3 months prior to the screening or planning to undergo any major surgery during the study.
* Presence or suspicion of ongoing of any serious infection.
* Human immunodeficiency virus (HIV) infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline in percent atheroma volume (PAV) | 52 weeks after treatment

SECONDARY OUTCOMES:
Change from the baseline in percent atheroma volume (PAV) | 24 weeks after treatment
Incidence of treatment-emergent adverse events (Safety and Tolerability) TEAEs and SAEs, and clinically significant changes in physical examination, vital signs, safety laboratory tests, and 12-lead ECG. | up to 14 days post the last dose of study drug

CONTACTS AND LOCATIONS:
Locations (4):
- The Lundquist Institute, Torrance, California, United States
- Australia (2):
  - Core Research Group Pty Ltd, Brisbane
  - Cognivus, Wahroonga
- The Zhongshan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
There is no such demand at present.